CLINICAL TRIAL: NCT00041795
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of Neotrofin to Treat Patients With Sensory or Motor Neuropathy Caused by Chemotherapy for Cancer
Brief Title: Neotrofin for Treatment of Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeoTherapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 082-2001-005
Record Dates: First submitted 2002-07-16; First posted 2002-07-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Peripheral Nervous System Diseases; Chemotherapy-Induced Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — 4-((3-(1,6-dihyro-6-oxo-9H-purin-9-yl)-1-oxopropyl)amino)benzoic acid

INTERVENTIONS:
Drug: leteprinim potassium (Neotrofin)

SUMMARY:
This study will assess the safety and efficacy of Neotrofin in treating the peripheral neuropathy that results from chemotherapy for cancer.

ELIGIBILITY:
* Patient must have diagnosis of cancer and be receiving or have received chemotherapy that has resulted in sensory or motor neuropathy.
* Sensory or motor neuropathy must be >/= grade 2 per Common Toxicity Criteria at baseline.
* In patients diagnosed with multiple myeloma, grade 1 sensory or motor neuropathy is acceptable.
* Patient must have normal hematological cell counts.
* Patient must have a life expectancy of >/= 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence St. Joseph Medical Center, Burbank, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Medical Center, New York, New York
  - The Sarah Cannon Cancer Center, Nashville, Tennessee

REFERENCES:
- [Background] Grundman M, Farlow M, Peavy G, Kim HT, Capparelli E, Schultz AN, Salmon DP, Ferris SH, Mobs R, Thomas RG, Schafer K, Campbell K, Hake AM, Schoos B, Thal LJ; Alzheimer's Disease Cooperative Study. A phase I study of AIT-082 in healthy elderly volunteers. J Mol Neurosci. 2002 Jun;18(3):283-93. doi: 10.1385/jmn:18:3:283. PMID 12059047
- [Background] Di Iorio P, Virgilio A, Giuliani P, Ballerini P, Vianale G, Middlemiss PJ, Rathbone MP, Ciccarelli R. AIT-082 is neuroprotective against kainate-induced neuronal injury in rats. Exp Neurol. 2001 Jun;169(2):392-9. doi: 10.1006/exnr.2001.7654. PMID 11358452
- [Background] Rathbone MP, Middlemiss PJ, Gysbers JW, Andrew C, Herman MA, Reed JK, Ciccarelli R, Di Iorio P, Caciagli F. Trophic effects of purines in neurons and glial cells. Prog Neurobiol. 1999 Dec;59(6):663-90. doi: 10.1016/s0301-0082(99)00017-9. PMID 10845757
- [Background] Middlemiss PJ, Glasky AJ, Rathbone MP, Werstuik E, Hindley S, Gysbers J. AIT-082, a unique purine derivative, enhances nerve growth factor mediated neurite outgrowth from PC12 cells. Neurosci Lett. 1995 Oct 20;199(2):131-4. doi: 10.1016/0304-3940(95)12029-4. PMID 8584241